CLINICAL TRIAL: NCT04465617
Title: Assessment of the Anterior Loop of the Inferior Alveolar Nerve in a Sample of Egyptian Population Using CBCT: An Observational Cross-Sectional Study
Brief Title: Assessment of the Anterior Loop of the IAN in a Sample of Egyptian Population Using CBCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Professor Hossam Kandil, Professor of Oral & Maxillofacial Radiology, Faculty of Dentistry, Cairo University
Other Study IDs: ORAD 7.1.1
Record Dates: First submitted 2020-06-28; First posted 2020-07-10 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-07

CONDITIONS: Mandibular Nerve
Keywords: Presence of the anterior loop of the mental nerve (branching from the inferior alveolar nerve) will be recorded & its length will be measured

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
in this study the prevalence & length of the anterior loop of the inferior alveolar nerve will be calculated and measured on retrospective CBCT patient's scans

DETAILED DESCRIPTION:
The proper knowledge of anatomical structures and their precise position is of a paramount importance for different dental specialties. The inferior alveolar nerve (IAN) canal is one of the most important anatomical landmarks in the mandible Shaban et al., 2017. By definition the inferior alveolar nerve (IAN) is a terminal division of the mandibular branch of the trigeminal nerve, it is confined within the mandibular canal and innervates all the mandibular teeth. The IAN initiates from the mandibular foramen and goes obliquely downward and forward in the ramus, and then horizontally within the body of the mandible. The IAN gives off the mental nerve, which exits the mandible through the mental foramen, supplying sensory branches to the chin, lower lip, mucous membranes and the gingiva; from the midline to about the second premolar region. It then continues its path anteriorly and turn into the mandibular incisive nerve, which innervates the mandibular canines and incisors Siddiqui et al. 2018. Before leaving the mental foramen and branching into the incisive nerve, the IAN may continue anteriorly and form an anterior loop (Al). This anterior loop is the part where the IAN directs mesially and occlusally before reversing direction and coursing distally towards the mental foramen Ragu et al., 2019. During implant planning and other surgical procedures knowing the presence of the anterior loop and its length is very crucial to avoid its injury. Specially concerning implantology where the location of the mental foramen and anterior loop determines the most distal point for implant placement in the interforaminal area; in order to avoid any injury resulting in sensory disturbances in this area Panjnoush et al., 2016 Recently, several studies have been published discussing the prevalence and length measurement of the anterior loop in many populations. However, no published researches were done on the Egyptian population. Therefore, this study is designed to assess the presence of the anterior loop and its length in a sample of Egyptian population using CBCT.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans of adult Egyptian patients, males and females.
* CBCT scans with unilateral or bilateral anterior mandibles; with minimum 2 mm length distal to the mental foramen

Exclusion Criteria:

* CBCT images of poor quality or artifacts interfering with the assessment of the anterior loop of IAN.
* Scans showing any pathosis in the interforaminal area (tumor or impaction).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult Egyptian population including males & females
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the anterior loop | 1 month
  it will be measured using CBCT axial cuts (Ondemand 3D software)

SECONDARY OUTCOMES:
length of the anterior loop | 1 month
  Built in measuring tools (axial cuts) in Ondemand 3D software "MPR* module"
Mesial extension of the anterior loop | 1 month
  Cross-sectional cuts on Ondemand 3D software "DVR** module"

CONTACTS AND LOCATIONS:
Locations (1):
- Orascan, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT04465617/Prot_SAP_000.pdf